CLINICAL TRIAL: NCT00243425
Title: Patient-Centered Depression Care for African Americans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: Aetna, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HS013645 (AHRQ)
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2005-10-24 (Estimated); Status verified 2005-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder;; African Americans;; Disparities;; Quality Improvement;; Patient Centered Care;; Primary Care;; Patient-Physician Relationship;
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Procedure: Standard Quality Improvement
Procedure: Patient-centered Intervention

SUMMARY:
The investigators propose to answer the following research question: Does a multifaceted, culturally tailored intervention that focuses on the specific concerns and preferences of African American patients with depression and their primary care providers improve the processes and outcomes of care for African Americans to a greater degree than a standard state-of-the art depression intervention?

This study will determine whether two new educational programs can improve the care for depression in African Americans. These programs may include visits with a depression case manager and access to educational materials, such as a videotape, a calendar, pamphlets, and books. One program is a standard quality improvement program for depression that has been shown to be effective in most patients. The other program is similar, but has materials that focus more on the patient's specific culture, beliefs, values, and preferences.

DETAILED DESCRIPTION:
Several studies document underutilization of outpatient specialty mental health services by African Americans. However, African Americans with depression are just as likely as whites to receive care in primary care settings. Despite their use of primary care services, African American patients are less likely than whites to be recognized as depressed, offered pharmacotherapy, and to initiate or complete pharmacotherapy or psychotherapy for depression. Compared to whites, African American patients express stronger preferences for counseling and more negative attitudes toward antidepressant medication, the most common form of treatment of depression used by primary care physicians. African Americans are also more likely to see depression and its treatment through a spiritual or religious framework. Studies show that African Americans receive less optimal technical and interpersonal health care than whites for many conditions. Depression is a common chronic condition that results in substantial morbidity, functional disability, and resource use. Despite the proven efficacy of pharmacotherapy and psychotherapy for treatment of depression, the gap between research findings and clinical practice is wide for management of depression in primary care. Recent intervention work has shown that quality improvement strategies for depression in primary care are effective. Research also shows that cultural adaptations can improve adherence and retention in care for ethnic minority patients. We have created a patient-centered adaptation that includes many of the components of recent successful quality improvement interventions for depression in primary care. The proposed study compares a standard depression intervention for patients (delivered by a depression case manager) and physicians (review of guidelines and structured mental health consultation) to a patient-centered intervention for patients (incorporates patient activation, individual preferences, and cultural sensitivity) and physicians (incorporates participatory communication skills training with individualized feedback on interactive CD-ROM). Thirty physicians and 250 patients will be randomized to either the standard interventions or the culturally tailored interventions. The main hypothesis is that patients in the patient-centered, culturally tailored intervention group will have higher remission rates from depression and lower levels of depressive symptoms at 12 months than patients in the standard intervention care group. Secondary outcomes will include patient receipt of guideline concordant care, patient and physician satisfaction with care, patient-physician communication behaviors, patient and physician attitudes towards depression, and self-efficacy in managing depression. This study will add to knowledge about how to effectively engage African American patients in care of depression and serve as a prototype of how to incorporate patient-centeredness in programs to reduce racial and ethnic disparities in health care for common conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have experienced two weeks or more of depressed mood/ loss of interest in the past year
* Patients who have experienced one week or more of depressed mood or loss of interest in the past month
* Self defined race or ethnicity African American
* Able to give written consent

Exclusion Criteria:

* Current alcohol or drug abuse
* History of mania
* Grief reaction or bereavement within the past 2 months
* Pregnancy
* Life expectancy less than 1 year
* Non English speaking
* Current specialty mental health care (at least 2 visits in past 6 weeks and appt scheduled in future
* Plan to change health care or primary care Provider in next 12 months
* Active suicidal thoughts and plans
* Residing in US for less than 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Compare the effectiveness of a culturally tailored intervention with the effectiveness of a standard intervention by evaluating its impact on patient outcomes (remission of depression, depression symptom level, functional status) at 6 and 12 months.

SECONDARY OUTCOMES:
Evaluating intervention impact on processes of care (satisfaction of care, guideline concordant care, patient involvement in participatory decision making, communication skills) rated by patients and providers at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cooper, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Christiana Care Health Services, Wilmington, Delaware
  - Johns Hopkins Community Phsyicians, Baltimore, Maryland
  - Sinai Hospital, Baltimore, Maryland
  - Baltimore Medical Systems, Middlesex Health Center, Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland

REFERENCES:
- [Background] Kaplan SH, Greenfield S, Ware JE Jr. Assessing the effects of physician-patient interactions on the outcomes of chronic disease. Med Care. 1989 Mar;27(3 Suppl):S110-27. doi: 10.1097/00005650-198903001-00010. PMID 2646486
- [Background] Roter DL, Stewart M, Putnam SM, Lipkin M Jr, Stiles W, Inui TS. Communication patterns of primary care physicians. JAMA. 1997 Jan 22-29;277(4):350-6. PMID 9002500
- [Background] Gallo JJ, Marino S, Ford D, Anthony JC. Filters on the pathway to mental health care, II. Sociodemographic factors. Psychol Med. 1995 Nov;25(6):1149-60. doi: 10.1017/s0033291700033122. PMID 8637945
- [Background] Cooper-Patrick L, Crum RM, Ford DE. Characteristics of patients with major depression who received care in general medical and specialty mental health settings. Med Care. 1994 Jan;32(1):15-24. doi: 10.1097/00005650-199401000-00002. PMID 8277799
- [Background] Cooper-Patrick L, Gallo JJ, Powe NR, Steinwachs DM, Eaton WW, Ford DE. Mental health service utilization by African Americans and Whites: the Baltimore Epidemiologic Catchment Area Follow-Up. Med Care. 1999 Oct;37(10):1034-45. doi: 10.1097/00005650-199910000-00007. PMID 10524370
- [Background] Cooper LA, Gonzales JJ, Gallo JJ, Rost KM, Meredith LS, Rubenstein LV, Wang NY, Ford DE. The acceptability of treatment for depression among African-American, Hispanic, and white primary care patients. Med Care. 2003 Apr;41(4):479-89. doi: 10.1097/01.MLR.0000053228.58042.E4. PMID 12665712
- [Background] Cooper LA, Roter DL, Johnson RL, Ford DE, Steinwachs DM, Powe NR. Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med. 2003 Dec 2;139(11):907-15. doi: 10.7326/0003-4819-139-11-200312020-00009. PMID 14644893
- [Background] Cooper-Patrick L, Powe NR, Jenckes MW, Gonzales JJ, Levine DM, Ford DE. Identification of patient attitudes and preferences regarding treatment of depression. J Gen Intern Med. 1997 Jul;12(7):431-8. doi: 10.1046/j.1525-1497.1997.00075.x. PMID 9229282
- [Derived] Cooper LA, Ford DE, Ghods BK, Roter DL, Primm AB, Larson SM, Gill JM, Noronha GJ, Shaya EK, Wang NY. A cluster randomized trial of standard quality improvement versus patient-centered interventions to enhance depression care for African Americans in the primary care setting: study protocol NCT00243425. Implement Sci. 2010 Feb 23;5:18. doi: 10.1186/1748-5908-5-18. PMID 20178624